CLINICAL TRIAL: NCT04068805
Title: Developing Affective HeaLth to Improve Adherence to Health Behaviors in Diabetes (DAHLIA II)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Sponsor chose to terminate this study for commercial reasons.
Sponsor: Happify Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Users are randomly assigned between arms after completing baseline assessment and stay in that arm for the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive affect condition (Active Comparator): Participants use Happify and have the option to use a diabetes-specific track that focuses on building skills for greater happiness, reducing stress, and coping better with diabetes. Users may access a wide variety of 4-week programs and use them in any way they desire for the entire study period.
  Interventions: Behavioral: Happify
- Psychoeducation condition (Sham Comparator): Participants complete a series of quizzes and polls on Happify designed to engage them in thinking about well-being topics, but without giving any specific instructions for how to promote well-being. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify

INTERVENTIONS:
Behavioral: Happify — An online platform for conveying techniques from positive psychology, cognitive-behavioral therapy, and mindfulness-based stress reduction.

SUMMARY:
Participants will be randomly assigned to either a positive affect skills intervention or a psychoeducation control group and assessed with questionnaires before, during, and after the 8-week program, as well as at 3 months, 6 months, and 12 months after the end of the program.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either the Diabetes positive affect skills intervention or a psychoeducation control group. Both programs last 8 weeks and take place on a simplified research version of the Happify platform. Participants assigned to the diabetes positive affect program will have full access to Happify, with a track that focuses on building skills for greater happiness, reducing stress, and coping better with diabetes displayed as the feature track. Participants assigned to the psychoeducation (control) condition will be asked to complete a series of polls on various wellbeing topics, and then provided with some social comparison data about how their responses compared with the responses of other users, as well as information about why the well being topic is important. Participants will be asked to complete questionnaires before, during, and after the 8-week program as well as 3 months, 6 months and 12 months follow-up questionnaires after the program is complete, at which point study participation will end.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Type 2 Diabetes
* Elevated HbA1c levels (7 or greater)
* No prior experience on the Happify platform (new user registration)
* PHQ-8 score of 13 or higher
* US resident
* Under the care of a medical professional for the treatment of their diabetes
* Be willing and able to obtain HbA1c every 3 months

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Change in self-reported HbA1C level | Baseline, 3 weeks post-intervention (day 83), 3 weeks after 3-month post intervention (day 173), 3 weeks after 6 month post intervention (day 263), and 12 months post intervention (day 416)
  1-item self-reported measure of Hemoglobin A1C (HbA1C) level, "What was your most recent HbA1c level?"

SECONDARY OUTCOMES:
Change in Depression symptoms [PHQ-9 questionnaire] | Baseline, immediate post-intervention at 8 weeks, and at 3, 6, and 12 months post-intervention
  9-item measure of depressive symptoms scoring how often the participant has been bothered by each statement over the past 2 weeks from not at all (0) to nearly every day (3).
Change in Diabetes Regimen Adherence | From baseline up to 63 days, 7 days at 3 months post intervention (146-153), 7 days at 6 months post intervention (236-243), and 12 months post intervention (day 416-423)
  1-item measure on keeping up with diabetes regimen in the past 24 hours, asking "Which of the following activities in your diabetes regimen did you complete over the past 24 hours?"
Change in Perceived Stress [Perceived Stress Scale (PSS)] | Baseline, immediate post-intervention at 8 weeks, and at 3, 6, and 12 months post-intervention
  10-item measure of perceived stress scoring how often the participant felt stressed by each statement in the following month from never (0) to very often (4).
Change in diabetes self-care activities [Summary of Diabetes Self-Care Activities (SDSCA)] | Baseline, immediate post-intervention at 8 weeks, and at 3, 6, and 12 months post-intervention
  11-item measure of self-reported adherence to diabetes self-care activities, ex. "On how many of the last seven days did you participate in at least 30 minutes of physical activity?" with possible answers of 0 to 7 days for each question.
Change in positive affect [Patient-Reported Outcomes Measurement Information Systems - Positive Affect Subscale(PROMIS)] | Baseline, immediate post-intervention at 8 weeks, and at 3, 6, and 12 months post-intervention
  15-item measure of positive affect scoring participants on how often then felt each statement was true over the past 7 days from not at all (1) to very much (5)

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Boucher, PhD, Principal Investigator — Happify Inc.
Locations (1):
- Happify (an online platform -- study is entirely online), New York, New York, United States

REFERENCES:
- [Derived] Boucher E, Moskowitz JT, Kackloudis GM, Stafford JL, Kwok I, Parks AC. Immediate and Long-Term Effects of an 8-Week Digital Mental Health Intervention on Adults With Poorly Managed Type 2 Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Aug 4;9(8):e18578. doi: 10.2196/18578. PMID 32749998